CLINICAL TRIAL: NCT01575626
Title: The Effect of Different Sevoflurane Concentrations on Intraocular Pressure in Patients Undergoing Ocular Surgery Under General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: TASMC-12-IM-0011-CTIL
Record Dates: First submitted 2012-03-28; First posted 2012-04-11 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: IOP Changes Due to Anesthesia (Healthy Patients)
MeSH Terms: interventions — Sevoflurane

ARMS (4):
- first sevoflurane concentration (Active Comparator): patients will be given 3 different end-tidal sevoflurane concentrations in the following order: 0%, 7%, 4%
  Interventions: Drug: Sevoflurane
- second sevoflurane concentration (Active Comparator): patients will be given 3 different end-tidal sevoflurane concentrations in the following order: 4%, 7%, 0%
  Interventions: Drug: Sevoflurane
- third sevoflurane concentration (Active Comparator): patients will be given 3 different end-tidal sevoflurane concentrations in the following order: 7%, 4%, 0%
  Interventions: Drug: Sevoflurane
- Propofol (Active Comparator): General anesthesia will be induced using propofol (5 mcg/ml) administered by target controlled infusion (TCI - Schnider model).Following tracheal intubation, concentration of propofol will be decreased till 0.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — All active comparators of this study have the same intervention as mentioned ahead:
  First IOP measurement will be performed just before anesthesia induction. Standard general anesthesia will be induced using propofol (5 mcg/ml) administered by target controlled infusion (TCI - Schnider model),fentanyl and rocuronium according to standard protocol of general anesthesia. The second IOP measurement will be performed just before tracheal intubation.
  Following tracheal intubation, concentration of propofol will be decreased till 0 and anesthesia with sevoflurane will be started, followed by 3 more IOP measurements for different end-tidal sevoflurane concentrations (Consented patients will be randomly allocated to one of three groups as mentioned).
  Total of 5 IOP measurements. IOP will be measured by the ophthalmologist via both TonoPen XL and Schioz devices.

SUMMARY:
One important goal in anesthetic management during ocular surgery is to provide adequate control of intraocular pressure (IOP). An increase in IOP may be catastrophic in patients with glaucoma or a penetrating open-eye injury. There is an ongoing debate over the effect of anesthetic agents on the IOP. Anesthetic regimens in this surgical field commonly consist of short-acting anesthetic agents, such as propofol and sevoflurane, usually combined with short-acting analgesics, such as remifentanil. Both propofol and sevoflurane are known to reduce the IOP. To this end there is no data in the literature to support or disprove this finding.

Study Hypothesis Variations in the end-tidal sevoflurane concentrations have no significant effect on the IOP.

DETAILED DESCRIPTION:
One important goal in anesthetic management during ocular surgery is to provide adequate control of intraocular pressure (IOP). An increase in IOP may be catastrophic in patients with glaucoma or a penetrating open-eye injury. There is an ongoing debate over the effect of anesthetic agents on the IOP. Anesthetic regimens in this surgical field commonly consist of short-acting anesthetic agents, such as propofol and sevoflurane, usually combined with short-acting analgesics, such as remifentanil. Both propofol and sevoflurane are known to reduce the IOP. Previous studies have compared these two anesthetics protocols in order to determine which provides superior control of the IOP. Propofol produced significantly lower IOP measurements compared to sevoflurane (both combined with remifentanil), in cataract surgery, whereas in non-ophthalmic surgery propofol and sevoflurane caused a comparable decrease in IOP. Sevoflurane, an inhalational anesthetic, has a rapid onset of action faster recovery time and is also suitable for inhalation induction because it does not irritate the airway. A prospective randomized clinical trial compared the effects of ketamine and sevoflurane on IOP during the eight minutes after induction of anesthesia (in 2-minute intervals) in children with suspected or diagnosed glaucoma undergoing EUA. During these 8 minutes the IOP decreased significantly only in the sevoflurane group. This finding contradicted claims that measurements immediately after induction are relatively unaffected by anesthetics and suggested that variations in sevoflurane concentration do affect the IOP. Yoshitake et al showed that the remarkable reductions of IOP after inductions are probably caused by induction agents, suggesting that sevoflurane is a useful anesthetic for elderly patients receiving ophthalmic surgeries. To this end there is no data in the literature to support or disprove this finding.

Study Hypothesis Variations in the end-tidal sevoflurane concentrations have no significant effect on the IOP.

ELIGIBILITY:
Inclusion Criteria:

* The study will include both men and women over 18 years old undergoing elective surgery for strabismus correction or tear duct probing and irrigation under general anesthesia.

Exclusion Criteria:

* Patients with known allergies,
* adverse reaction or contraindication (of any other reason) to sevoflurane or remifentanil, or any other anesthetic drug,
* patients with pre-existing intra-ocular ophthalmic disease, or infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
effect of different end-tidal sevoflurane concentrations on the IOP | 1 year
  To assess the effect of different end-tidal sevoflurane concentrations on the IOP in patients undergoing extraocular procedures, i.e. strabismus correction and tear duct probing and irrigation under general anesthesia.

SECONDARY OUTCOMES:
propofol vs. sevoflurane on IOP | 1 year
  To compare the influence of propofol vs. sevoflurane on IOP

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel